CLINICAL TRIAL: NCT01648296
Title: Measurements of Myocardial Fatty Acid Metabolism With PET and [F-18]FluorbetaOx in Humans With Heart Failure With and Without Diabetes: Comparison With [C-11]Palmitate
Brief Title: Fatty Acid Radiotracer Comparison Study in Heart Failure Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IND113344; IRB#201208087 (Other: Human Research Protection Office at Washington University)
Record Dates: First submitted 2012-07-11; First posted 2012-07-24 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure; Obesity; Type 2 Diabetes Mellitus; Health Normal Volunteer Subjects
Keywords: Heart Failure; Obesity; Type 2 Diabetes Mellitus; Health Normal Volunteer Subjects
MeSH Terms: conditions — Heart Failure; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Dosimetry Group (Experimental): A total of 12 subjects will receive a single intravenous injection of[18F]FluorbetaOx followed by PET-CT imaging. Four normal healthy volunteer subjects and 8 subjects with or without Type 2 Diabetes Mellitus with Chronic Dilated Cardiomyopathy.
  Interventions: Drug: [18F]FluorbetaOx
- Kinetic Dynamic Group (Experimental): A total of 38 subjects will receive a single intravenous injection of [18F]FluorbetaOx, [11C]Palmitate, and [15O]Water followed by PET-CT imaging. Ten normal healthy volunteer subjects and 28 subjects with or without Type 2 Diabetes Mellitus of which 18 subjects will have Chronic Dilated Cardiomyopathy and 10 obese subjects with a Body Mass Index of ≥ 30kg/m2.
  Interventions: Drug: [18F]FluorbetaOx

INTERVENTIONS:
Drug: [18F]FluorbetaOx — Fluorine 18-labeled FluorbetaOx
  Other Names: IND #113344

SUMMARY:
A single center, open-label baseline controlled imaging study to designed to assess whether Positron Emission Tomography (PET) measurements of myocardial Fatty Acid (FA) metabolism performed with [18F]FluorbetaOx correlates with measurements using [11C]palmitate. This study involves the investigational use of a PET radioactive tracer, fluorine-18 radiolabeled fatty acid analog, [18F]FluorbetaOx designed to measure beta oxidation of fatty acids in the myocardium. The investigators propose to evaluate the feasibility of the method in heart failure patients with dilated non-ischemic cardiomyopathy (DCM) with or without type-2 diabetes mellitus (T2DM) and obese subjects (Body Mass Index of ≥ 30kg/m2) with or without T2DM and normal healthy subjects to provide a wide range of perturbations in myocardial FA metabolism.

Specific objectives include:

1. To assess the diagnostic quality of [18F]FluorbetaOx PET images and kinetics at the proposed 10 millicurie (mCi) dose.
2. To quantitatively determine the relationship between PET measurements of myocardial FA metabolism obtained with [18F]FluorbetaOx and those using [11C]Palmitate.
3. To calculate human dosimetry based on the human biodistribution of [18F]FluorbetaOx.
4. Correlate measurements of myocardial FA metabolism with changes in left ventricular (LV)structure and function performed on a clinically indicated echocardiography at 6-9 months after imaging.

DETAILED DESCRIPTION:
PET imaging will be broken down into 2 groups of subjects (dosimetry and kinetic dynamic imaging/[11C]palmitate comparison) with entry into these groups will occur simultaneously. All PET imaging will be performed with a Siemens Biograph 40 PET-CT scanner. All patients will undergo routine clinical evaluation as dictated by the treating heart failure cardiologist. The results of the PET studies will not be provided to the patient or the treating cardiologist unless, in the judgment of the Principal Investigator, the images demonstrate an unsuspected abnormality that may warrant further evaluation. Subjects will be instructed not to eat after midnight the night before the study. However, patients will be instructed to continue their heart failure and diabetic medical regimens. The morning of their PET study, subjects will have two intravenous catheters placed. One will be placed in each arm for the purpose of administering radioactive tracers ([15O]Water, [11C]Palmitate, and [18F]FluorbetaOx), drawing blood samples for safety laboratory analysis. Urine samples will be obtained along with an Electrocardiogram (ECG) and vital signs. A follow-up telephone contact will be done 2-3 days post imaging study to capture unanticipated and serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years of age inclusive, at the time of signing the informed consent
* Chronic dilated cardiomyopathy of non-ischemic origin
* New York Heart Association (NYHA)Class II/III heart failure for a minimum of 6 months prior to enrollment
* Heart Failure patients with Left Ventricular Ejection Fracture less than or equal to 35%
* Obesity defined as Body Mass Index of ≥ 30kg/m2
* Type 2 Diabetes Mellitus based on standard American Diabetes Association (ADA) criteria
* Capable of giving informed consent
* Not currently pregnant or nursing: Female subjects must be either: surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (cessation of menses for more than 1 year), or of childbearing potential for whom a urine pregnancy test (with the test performed within the 24 hour period immediately prior to administration of [18F] FluorbetaOx is negative

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A recent positive pre-study drug/alcohol screen noted in medical records
* Pregnant females as determined by positive (serum or urine) human chorionic gonadotropin(hCG) test at screening or prior to dosing
* Lactating females
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated
* History of a psychiatric disorder that will affect the subject's ability to participate in the study
* Restrictive, obstructive, or infiltrative cardiomyopathy; pericardial disease; uncorrected thyroid disease (TSH) noted in medical records
* History of clinically significant coronary artery disease (CAD)including (prior (ST) elevation myocardial infarction, presence of ≥ 50% obstruction of a major coronary artery, and presence of angina)
* Contraindications to PET scanning (i.e., inability to lie flat with arms over head for up to 1½ hours; claustrophobia; current participation in research studies involving radiation exposure such that the total research-related radiation dose to the subject in any given year would exceed the Code of Federal Regulation limits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09-13 (Actual); Primary Completion 2014-06-04 (Actual); Study Completion 2014-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Gropler, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dosimetry Group | Kinetic Dynamic Group
Started | 11 | 17
Completed | 11 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dosimetry Group | Kinetic Dynamic Group | Total
Number analyzed (Participants) | 11 | 17 | 28
Age, Continuous [Median (Full Range); unit: years] | 46.5 [18 to 75] | 46.5 [18 to 75] | 46.5 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 5 | 9 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is to Determine if PET/CT Measurements of Myocardial FA Metabolism Performed With [18F]FluorbetaOx Correlated With Those Performed With [11C]Palmitate and Calculation of Human Dosimetry.
Description: The values in the table represent the number of participants, specifically Dosimetry and Kinetic patients and that is how the primary endpoint is arrived at. This is how the primary endpoint is determined through PET/CT measurements of Myocardial FA metabolism with F-18 Florbeta Ox.
  The data intended for this Outcome Measure use PET/CT images to visualize the amount of myocardial FA metabolism appears with the radio tracer, Florbeta Ox.
Time Frame: 24-72 hrs
Population: The PI has left the institution, all efforts to locate this data have been exhausted and it therefore cannot be reported
Arm/Group | Dosimetry Group | Kinetic Dynamic Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Determine Human Dosimetry Based on the Human Biodistribution of [18F](+/-)NOS in Both Normal Healthy Volunteers and Dilated Non-ischemic Cardiomyopathy Patients.
Description: A total of 0 subjects (Four normal healthy volunteer subjects and0 subjects with or without Type 2 Diabetes Mellitus with Chronic Dilated Cardiomyopathy)will receive a single intravenous injection of 10 mCi of[18F]FluorbetaOx followed by PET-CT imaging at two separate time points.
  The difference between primary Outcome and the secondary outcome are the patients themselves. Florbeta Ox was measured in normal healthy volunteers and in non-ischemic cardiomyopathy patients through PET/CT image visualization.
Time Frame: 2-3 days post [18F]FluorbetaOx injection
Population: The PI has left the institution, and all efforts to locate this data have been exhausted and it therefore cannot be reported.
Groups:
- Dosimetry Group: A total of 0 subjects will receive a single intravenous injection of[18F]FluorbetaOx followed by PET-CT imaging. Four normal healthy volunteer subjects and 8 subjects with or without Type 2 Diabetes Mellitus with Chronic Dilated Cardiomyopathy.
  [18F]FluorbetaOx: Fluorine 18-labeled FluorbetaOx
- Kinetic Dynamic Group: A total of 0subjects will receive a single intravenous injection of [18F]FluorbetaOx, [11C]Palmitate, and [15O]Water followed by PET-CT imaging. Ten normal healthy volunteer subjects and 28 subjects with or without Type 2 Diabetes Mellitus of which 18 subjects will have Chronic Dilated Cardiomyopathy and 10 obese subjects with a Body Mass Index of ≥ 30kg/m2.
  [18F]FluorbetaOx: Fluorine 18-labeled FluorbetaOx
Arm/Group | Dosimetry Group | Kinetic Dynamic Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Dosimetry Group | Kinetic Dynamic Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/17
Other Adverse Events (participants affected / at risk) | 0/11 | 0/17

LIMITATIONS AND CAVEATS:
There are no limitations and caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes